CLINICAL TRIAL: NCT00365950
Title: Clinical Trial of Two Durations of Warfarin Therapy in the Treatment of Deep Vein Thrombosis and/or Pulmonary Embolism
Brief Title: 3 Months' Versus 6 Months' Anticoagulation in Patients With DVT and/or PE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: British Thoracic Society (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTS DVT/PE Study
Record Dates: First submitted 2006-08-17; First posted 2006-08-18 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2004-01

CONDITIONS: Deep Vein Thrombosis; Pulmonary Embolism; Deep Vein Thrombosis With Pulmonary Embolism
Keywords: Duration of anticoagulation; Deep vein thrombosis and/or pulmonary embolism
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism

INTERVENTIONS:
Drug: Duration of anticoagulation
Drug: Warfarin duration

SUMMARY:
To determine whether 3 months' anticoagulation is as good as or better than 6 months' for the treatment of DVT/PE

DETAILED DESCRIPTION:
Multi-centre trial involving 46 hospitals in the United Kingdom, with patients entered by 137 Consultant Physicians. Consenting patients were randomised in a central office to either 3 months' or 6 months' anticoagulation. Information on progress of the patients was requested by the co-ordinating office at 3 months, 6 months and 12 months. Outcomes were measured as death from DVT/PE, non-fatal extensions or recurrences of DVT/PE and major haemorrhages during and after anticoagulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or more with suspected or proven DVT/PE whom the clinician intended to anticoagulate.

Exclusion Criteria:

* DVT/PE severe enough to require thrombolysis or pulmonary embolectomy.
* DVT/PE in the preceding 3 years.
* Neoplasia diagnosed/treated within previous 3 years.
* Pregnancy.
* Known major thrombophilias.
* Prolonged or continuous immobility or confinement to bed.
* Previous allergy to heparin or warfarin.
* Requirement for long-term anticoagulation.
* Inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400
Dates: Start 1999-09; Study Completion 2003-12

PRIMARY OUTCOMES:
Death due to DVT/PE
Failures of resolution, extension or recurrence of DVT and/or PE during and after treatment.
Number of major haemorrhages.

SECONDARY OUTCOMES:
Comparison of length of Hospital stay between those given unfractionated heparin and those given low molecular weight heparin.

CONTACTS AND LOCATIONS:
Overall Officials: Aziz Sheikh, MD,FRCGP, Study Chair — Research Committee of the British Thoracic Society
Locations (2):
- United Kingdom (2):
  - Department of Chest Medicine, Llandough Hospital, Cardiff, Wales
  - Department of Chest Medicine, Llandough Hospital,, Cardiff, Wales

REFERENCES:
- [Derived] Campbell IA, Bentley DP, Prescott RJ, Routledge PA, Shetty HG, Williamson IJ. Anticoagulation for three versus six months in patients with deep vein thrombosis or pulmonary embolism, or both: randomised trial. BMJ. 2007 Mar 31;334(7595):674. doi: 10.1136/bmj.39098.583356.55. Epub 2007 Feb 8. PMID 17289685